CLINICAL TRIAL: NCT02632630
Title: Nutrition Supplementation in Hospitalized Patients: A Randomized Controlled Trial
Brief Title: Nutrition Supplementation in Hospitalized Patients
Acronym: NutriSuP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Academic Medical Organization of Southwestern Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: INN15-007
Record Dates: First submitted 2015-12-03; First posted 2015-12-17 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Malnutrition
Keywords: Peripheral Parenteral Nutrition; Oral nutritional supplementation; Acute Care hospitals
MeSH Terms: conditions — Malnutrition | interventions — Glucose; Crystalloid Solutions; Saline Solution; Ringer's Lactate; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Amino Acids w/Electrolytes in Dextrose (Active Comparator): Peripheral parenteral nutrition (PPN)
  Interventions: Drug: Amino Acids w/Electrolytes in Dextrose
- Ensure product (Active Comparator): Calorie and protein dense oral nutritional supplement for patients with elevated nutritional needs.
  Interventions: Dietary Supplement: Ensure product
- Crystalloid solutions (Active Comparator): Standard care intravenous maintenance fluids.
  Interventions: Drug: Crystalloid solutions
- Oral nutritional supplementation (Active Comparator): Nutrient-enhanced drink products that provide macronutrients and micronutrients with the aim of increasing oral nutritional intake.
  Interventions: Dietary Supplement: Oral nutritional supplementation

INTERVENTIONS:
Drug: Amino Acids w/Electrolytes in Dextrose — Patients will receive peripheral parenteral nutrition to a maximum of 2L/day (with a minimum rate of 45mL/hour and a maximum rate of 85mL/hour) of pre-packaged Peri-OLIMEL 2.5% E. The PPN will be administered in place of their maintenance crystalloid solution, and will be adjusted or stopped as clinically indicated by the attending medical team., for up to 5 days of hospitalization or until discharge, whichever is sooner.
  Other Names: Peri-OLIMEL 2.5% E (Baxter)
  Arms: Amino Acids w/Electrolytes in Dextrose
Dietary Supplement: Ensure product — Patients will receive one package of Ensure two times daily in hospital. At discharge, patients randomized to receive Ensure will be provided with 28 packages of Ensure with instructions to attempt to consume 1 package per day.
  Arms: Ensure product
Drug: Crystalloid solutions — Standard care intravenous maintenance fluid administration for up to 5 days of hospitalization or until discharge, whichever is sooner.
  Other Names: normal saline, dextrose, lactated Ringer's
  Arms: Crystalloid solutions
Dietary Supplement: Oral nutritional supplementation — Standard of care oral nutritional supplementation is determined by the clinician. A dietitian may also be involved.
  Arms: Oral nutritional supplementation

SUMMARY:
Patients with severe malnutrition risk are 7.4 times more likely to die in hospital than well-nourished patients, and carry a 30-day readmission rate of >46%. Although malnutrition is common and is associated with extremely poor outcomes, it is neglected and undertreated. This is a randomized controlled pilot trial to rapidly identify at-risk hospitalized medical patients, and then provide nutritional supplementation in hospital and after discharge for 28 days. In select at-risk patients, 5 days of nutrition delivered through a peripheral vein will be used in addition to oral nutritional supplementation.

DETAILED DESCRIPTION:
In this pilot trial, the feasibility of the trial protocol will be established in two centres in Canada. Patients at high risk of malnutrition will be identified within 48 hours of hospital admission using Subjective Global Assessment criteria. Patients will be randomized in a factorial design fashion via a centralized, internet-based randomization protocol to one of the following arms:

1. Peripheral parenteral nutrition and enhanced oral supplementation;
2. Peripheral parenteral nutrition and standard care for oral supplementation;
3. Standard care for parenteral fluid administration and enhanced oral supplementation;
4. Standard care for parenteral fluid administration and standard of care for oral supplementation.

Peripheral parenteral nutrition (PPN) is intravenous nutrition consisting of dextrose, amino acids, fat, and electrolytes through a peripheral vein. Peri-OLIMEL 2.5% E, parenteral solution (Baxter) will be administered in this study. Patients will be randomized to PPN vs. standard care intravenous maintenance fluid administration for up to 5 days of hospitalization or until discharge, whichever is sooner. The PPN will be administered in place of their maintenance crystalloid solution, and will be adjusted or stopped as clinically indicated by the attending medical team.

If there is no maintenance crystalloid fluid administration, the parenteral nutrition solution will be administered at a rate of 0.85mL/kg/hour.

The minimum infusion rate will be 45 mL per hour (for participants who weigh 53 kg or less). The minimum infusion rate would provide a supplementation of 1,080 kcal/day.

The maximum infusion rate will be 85 mL/hour (for participants who weigh 100 kg or more). The maximum infusion rate would provide a supplementation of 2,040 kcal/day.

The PPN solution has a low osmolarity (< 900 mOsm) to reduce risk of phlebitis (Peri-OLIMEL 2.5% E is760mOsm). The use of PPN, compared to total parenteral nutrition (TPN) offers safety advantages. PPN avoids cost and complication of central line placement, avoids line sepsis and reduces the likelihood re-feeding syndrome [30-32]. Peri-OLIMEL 2.5% E contains lipids and electrolytes further reducing the likelihood of vein irritation and refeeding syndrome. All patients will be monitored closely and patients with uncontrolled blood sugars will be excluded.

Patients randomized to Oral Nutritional Supplementation (ONS) will receive standard menu or standard menu plus oral nutritional supplements. The investigators will provide patients with one package of ONS (Resource 2.0 - 237 mL, 474 calories; or similar product) two times daily in hospital. Although the patient will be encouraged, they will not be required to consume all of the oral supplementation product. Upon discharge, patients will be provided with ONS product to take home.

All participants will be monitored daily in hospital. After discharge, the investigators will follow up with the participant at a 30-day follow-up clinic visit, to collect data regarding clinical outcomes, quality of life, physical function, and nutrition-related variables.

This pilot study will establish the feasibility of a paradigm-changing protocol that will rapidly identify and aggressively treat malnutrition in hospitalized patients, with the goal of improving function, quality of life, healthcare utilization, and reducing the risk of adverse clinical events.

ELIGIBILITY:
Inclusion Criteria:

* Subjective Global Assessment (SGA) category B or C.
* Have been hospitalized for less than 48 hours.

Exclusion Criteria:

* Have an allergy or intolerance to any component of the oral supplement or parenteral nutrition.
* Have a contraindication to administration of IV fluid (i.e. are in volume overloaded state, are being given IV furosemide).
* Are currently suffering from refeeding syndrome.
* Have a pre-existing medical condition that prevents oral intake of full fluids.
* Have a diagnosis or suspicion of septic shock.
* Have an expected length of stay of less than 48 hours from the time of assessment.
* Have a current diagnosis of diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Successful participant recruitment | 12 months
  This pilot study will demonstrate feasibility of recruitment if investigators are able to recruit 100 participants over 12 months. A total recruitment of 15 patients/month is considered as reasonable given the high numbers of competing studies, missed patients, and consent failure rates.

SECONDARY OUTCOMES:
Adherence to treatment | 30 days
  Adherence to the study treatments will be defined as ≥90% of prescribed intervention being administered across all patients. Preliminary estimates of non-administration of the trial intervention are needed, along with strategies that maximize exposure to the intervention.
Number of participants to experience clinical re-feeding syndrome. | 30 days
  It is expected that some participants will experience metabolic electrolyte abnormalities related to initiation of feeding requiring electrolyte and fluid replacement but it is expected that clinical re-feeding syndrome characterized by cardiac, pulmonary, neurological abnormalities will be absent; an opinion informed by the investigators' recent systematic review.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Rahman, MD, FRCPC, Principal Investigator — St. Joseph's Health Care
Locations (1):
- LHSC-University Hospital, London, Ontario, Canada

REFERENCES:
- [Derived] Mrkobrada M, Patel A, Chakroborty A, Handsor S, Armstrong D, Rahman A. NutriSup-PPN: A pilot randomized control trial of oral nutritional supplementation (ONS) and peripheral parenteral nutrition (PPN) in canadian, malnourished, hospitalized patients. Clin Nutr ESPEN. 2023 Feb;53:107-112. doi: 10.1016/j.clnesp.2022.04.008. Epub 2022 Apr 23. PMID 36657900